CLINICAL TRIAL: NCT06965647
Title: The Effect of Partner-Conducted Fetal Heart Sound Measurement on Maternal-Paternal Expectations and Maternal-Paternal Attachment: An Experimental Study
Brief Title: Effect of Partner-Conducted Fetal Heart Sound Measurement on Maternal and Paternal Attachment
Acronym: FHS-ATTACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Kader ATABEY, Research Assistant, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10576553
Record Dates: First submitted 2024-06-18; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-12

CONDITIONS: Prenatal Attachment, Maternal Expectations, Paternal Involvement
Keywords: motherhood, fatherhood, prenatal attachment, partner involvement, fetal heart sound, parental expectations

STUDY DESIGN:
Intervention Model Description: Randomized controlled design with parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Couples who met the inclusion criteria were invited from Hasköy Family Health Center. Based on national prenatal care guidelines, two sessions were scheduled at 28-32 weeks and 33-38 weeks of gestation. Fathers were trained on Leopold maneuvers and fetal heart sound measurement. Under midwife supervision, fathers performed Leopold maneuvers and fetal heart sound measurements using a Doppler device. The intervention was applied twice.
  Interventions: Behavioral: Partner-Conducted Fetal Heart Sound Measurement
- Control Group (No Intervention): Couples in the control group received standard prenatal follow-up. At 28-32 and 33-38 weeks, data were collected using the same tools without any intervention. During routine visits, the fetal heart sound measurement and Leopold maneuvers were performed by the midwife as part of standard care.

INTERVENTIONS:
Behavioral: Partner-Conducted Fetal Heart Sound Measurement — Expectant fathers in the intervention group were trained in basic Leopold maneuvers and fetal heart sound measurement using a Doppler device. Under the supervision of a midwife, fathers located the fetus's back, applied gel, and measured the heart sound during prenatal visits at 28-32 and 33-38 weeks of gestation.
  Arms: Intervention Group

SUMMARY:
This randomized controlled study aims to evaluate the effect of fetal heart sound (FHS) measurement performed by the partner on prenatal maternal and paternal expectations and attachment levels. A total of 120 couples (60 intervention, 60 control) participated in the study.

DETAILED DESCRIPTION:
This experimental study was conducted to determine the effect of partner-conducted fetal heart sound (FHS) measurement on prenatal maternal and paternal expectations and attachment. The study included 120 couples (60 intervention, 60 control) whose pregnancies were between 28 and 38 weeks, and who were registered at Hasköy Family Health Center in Muş, Turkey. In the intervention group, the father was trained in Leopold maneuvers and performed the FHS measurement twice - once during 28-32 weeks and again during 33-38 weeks of gestation. Data collection tools included the Prenatal Maternity Expectations Scale, Prenatal Paternity Expectations Scale, Prenatal Attachment Inventory, and the Paternal Antenatal Attachment Scale. Data were collected before the first FHS measurement (pre-test) and after the second (post-test). The control group received standard prenatal monitoring by healthcare staff without involving the partner. The study was approved by the Malatya Clinical Research Ethics Committee (Approval No: 2022/3968).

ELIGIBILITY:
- Inclusion Criteria: Women between 28 and 38 weeks of gestation

* Age between 18 and 45 years
* Ability to read and write
* No diagnosed psychiatric illness
* Healthy pregnancy
* Attending prenatal visits with their partner

Exclusion Criteria:

* Women with diagnosed psychiatric conditions
* Couples unwilling to participate
* Incomplete data forms
* Those who moved out of the study area during follow-up
* Women without their partners during visits

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Prenatal Paternal Attachment Level | From 28-38 weeks of gestation (approximately 10 weeks)
  Change in paternal attachment scores, measured using the Prenatal Paternal Attachment Scale (PPAS), before and after partner-conducted fetal heart sound measurement.

SECONDARY OUTCOMES:
Prenatal Maternal Attachment Level | From 28-38 weeks of gestation (approximately 10 weeks)
  Change in maternal attachment scores, measured using the Prenatal Attachment Inventory (PAI), before and after the intervention.
Parental Expectations (Mother and Father) | From 28-38 weeks of gestation (approximately 10 weeks)
  Change in maternal and paternal expectations measured using validated Maternity and Paternity Expectation Scales before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- İnönü üniversitesi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD).